CLINICAL TRIAL: NCT02200172
Title: The Preventative Role of Exogenous Melatonin Administration in Patients With Advanced Cancer Who Are at Risk of Delirium: a Feasibility Study Prior to a Larger Randomized Controlled Trial
Brief Title: The Preventative Role of Exogenous Melatonin Administration in Patients With Advanced Cancer Who Are at Risk of Delirium: a Feasibility Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BRI-MELAT-2013
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: Cancer; Melatonin; Delirium; Feasibility Studies; Palliative Care
MeSH Terms: conditions — Neoplasms; Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator): A single daily sublingually administered tablet of 3mg non-animal synthetic source melatonin (immediate-release) at 21.00 hours (±1 hour), starting on Study Day 1 and stopping on Study Day 28 of admission or earlier in the event of death or discharge.
  Interventions: Other: Melatonin
- Placebo (Placebo Comparator): A single daily sublingually administered tablet of placebo at 21.00 hours (±1 hour), starting on Study Day 1 and stopping on Study Day 28 of admission or earlier in the event of death or discharge.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Melatonin — Sublingual 3mg non-animal synthetic source melatonin daily at 21.00 hours (±1 hour).
  Arms: Melatonin
Other: Placebo
  Other Names: Sublingual placebo daily at 21.00 hours (±1 hour).
  Arms: Placebo

SUMMARY:
The purpose of this feasibility study is to inform a larger randomized, placebo-controlled, double blind, parallel-group, single-centre trial of an oral, daily administered single dose of melatonin to prevent delirium in patients with advanced cancer.

DETAILED DESCRIPTION:
Delirium is a very common and distressing neuropsychiatric syndrome in palliative care and a variety of other settings. It is associated with increases in morbidity, mortality, health care costs and most importantly in levels of patient and family distress. Inpatient palliative care is delivered in stand-alone hospice units and increasingly in designated units in acute care hospitals, where delirium occurrence rates of over 80% have been reported in the last hours and days before death. Most patients in these units have a cancer diagnosis. Given the increasing elderly proportion of the population, and that cancer is predominantly a disease of the elderly, there is a pivotal need to develop primary, secondary and tertiary preventative strategies for delirium in these patients.

Although sleep-wake cycle disturbance is not a core diagnostic criterion for delirium, studies of delirium in cancer patients have reported occurrence rates of 75-100%. This most likely reflects a circadian rhythm disturbance. Recent research suggests that giving melatonin to patients who are admitted to hospital may prevent them from developing delirium.

This feasibility study aims to inform a larger randomized, placebo-controlled, double blind, parallel-group, single-centre trial of an oral, daily administered single dose of melatonin to prevent delirium in patients with advanced cancer.

The study will be conducted on the 31-bed Palliative Care Unit (PCU), a university teaching unit, at Bruyère Continuing Care. The intervention consists of a single daily sublingually administered tablet of either 3mg non-animal synthetic source or placebo at 21.00 hours (±1 hour), starting on study day 1 and stopping on study day 28 of admission or earlier in the event of death or discharge. The study drug will be discontinued immediately if incident delirium occurs before day 28.

Throughout the trial, multiple dimensions of feasibility will be evaluated such as recruitment, retention and acceptability of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years
* Cancer diagnosis
* Admitted to Palliative Care Unit
* English speaking
* Cognitive capacity to give informed consent or substitute decision maker is accessible to provide consent
* Palliative Performance Scale ≥ 30% at the time of consent

Exclusion Criteria:

* Delirium present on admission (assessed clinically with the CAM)
* Known psychotic disorder other than dementia
* Inability to take medications sublingually or via gastrostomy tube
* Known allergy to melatonin or placebo content
* Use of melatonin within the two weeks preceding admission
* Patient on warfarin treatment or other oral anticoagulant
* Communication problems that cannot be accommodated, including deafness, tracheostomy, aphasia, dysarthria or emotional distress
* On other investigational agents or treatments
* Pregnancy or lactation
* Severe visual impairment or designated legally blind
* Immunosuppressant medication use in the context of autoimmune disease or post organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time to first onset of delirium for participants receiving active comparator versus placebo | 8 months
  Preliminary data will help determine the appropriateness of this outcome measure in a larger trial.
Number of times the blinding on the trial product is broken. | 8 months
  This number will indicate any further need for research team training.
Recruitment and retention rates | 8 months
  Recruitment and retention rates will determine if a larger trial with the same design will allow for a sufficient number of participants.
Frequency of protocol violation | 8 months
  The frequency of protocol violations will indicate if a larger trial with the same design can be implemented in a palliative care setting or require modification.
Number of unsolicited positive versus negative comments from participants, families, and Palliative Care Unit staff | 8 months
  Comments that are voluntarily provided will show whether the trial is acceptable to participants, families, Palliative Care Unit staff.

SECONDARY OUTCOMES:
Predisposing and precipitating risks form completion rate | 8 months
  Predisposing and precipitating factors will be collected on trial forms throughout the trial. The feasibility of collecting this data on the Palliative Care Unit will be measured by form completion rates.
Number of participants with serious adverse events related to the active comparator | Participants will be followed for the duration of trial product administration plus 2 days for an expected total of 30 days
  To assess the safety of the proposed intervention in this palliative care population will be assessed on an ongoing basis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lawlor, MB, MMedSc, Principal Investigator — Clinician Scientist, Bruyère Research Institute; Medical Director, Bruyère Continuing Care
Locations (1):
- Bruyère Continuing Care, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Hanania M, Kitain E. Melatonin for treatment and prevention of postoperative delirium. Anesth Analg. 2002 Feb;94(2):338-9, table of contents. doi: 10.1097/00000539-200202000-00019. PMID 11812694
- [Background] Al-Aama T, Brymer C, Gutmanis I, Woolmore-Goodwin SM, Esbaugh J, Dasgupta M. Melatonin decreases delirium in elderly patients: a randomized, placebo-controlled trial. Int J Geriatr Psychiatry. 2011 Jul;26(7):687-94. doi: 10.1002/gps.2582. Epub 2010 Sep 15. PMID 20845391
- [Background] Hagen NA, Biondo PD, Brasher PM, Stiles CR. Formal feasibility studies in palliative care: why they are important and how to conduct them. J Pain Symptom Manage. 2011 Aug;42(2):278-89. doi: 10.1016/j.jpainsymman.2010.11.015. Epub 2011 Mar 27. PMID 21444184
- [Background] Siddiqi N, Stockdale R, Britton AM, Holmes J. Interventions for preventing delirium in hospitalised patients. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD005563. doi: 10.1002/14651858.CD005563.pub2. PMID 17443600
- [Background] Tabet N, Howard R. Pharmacological treatment for the prevention of delirium: review of current evidence. Int J Geriatr Psychiatry. 2009 Oct;24(10):1037-44. doi: 10.1002/gps.2220. PMID 19226527
- [Background] Agar M, Lawlor P. Delirium in cancer patients: a focus on treatment-induced psychopathology. Curr Opin Oncol. 2008 Jul;20(4):360-6. doi: 10.1097/CCO.0b013e328302167d. PMID 18525328
- [Background] Lawlor PG, Fainsinger RL, Bruera ED. Delirium at the end of life: critical issues in clinical practice and research. JAMA. 2000 Nov 15;284(19):2427-9. doi: 10.1001/jama.284.19.2427. No abstract available. PMID 11074759
- [Background] Miyazaki T, Kuwano H, Kato H, Ando H, Kimura H, Inose T, Ohno T, Suzuki M, Nakajima M, Manda R, Fukuchi M, Tsukada K. Correlation between serum melatonin circadian rhythm and intensive care unit psychosis after thoracic esophagectomy. Surgery. 2003 Jun;133(6):662-8. doi: 10.1067/msy.2003.149. PMID 12796735
- [Background] Olofsson K, Alling C, Lundberg D, Malmros C. Abolished circadian rhythm of melatonin secretion in sedated and artificially ventilated intensive care patients. Acta Anaesthesiol Scand. 2004 Jul;48(6):679-84. doi: 10.1111/j.0001-5172.2004.00401.x. PMID 15196098
- [Background] de Jonghe A, van Munster BC, van Oosten HE, Goslings JC, Kloen P, van Rees C, Wolvius R, van Velde R, Levi MM, Korevaar JC, de Rooij SE; Amsterdam Delirium Study group. The effects of melatonin versus placebo on delirium in hip fracture patients: study protocol of a randomised, placebo-controlled, double blind trial. BMC Geriatr. 2011 Jul 5;11:34. doi: 10.1186/1471-2318-11-34. PMID 21729284
- [Background] de Jonghe A, Korevaar JC, van Munster BC, de Rooij SE. Effectiveness of melatonin treatment on circadian rhythm disturbances in dementia. Are there implications for delirium? A systematic review. Int J Geriatr Psychiatry. 2010 Dec;25(12):1201-8. doi: 10.1002/gps.2454. PMID 21086534
- [Derived] Lawlor PG, McNamara-Kilian MT, MacDonald AR, Momoli F, Tierney S, Lacaze-Masmonteil N, Dasgupta M, Agar M, Pereira JL, Currow DC, Bush SH. Melatonin to prevent delirium in patients with advanced cancer: a double blind, parallel, randomized, controlled, feasibility trial. BMC Palliat Care. 2020 Oct 21;19(1):163. doi: 10.1186/s12904-020-00669-z. PMID 33087111
- [Derived] Bush SH, Lacaze-Masmonteil N, McNamara-Kilian MT, MacDonald AR, Tierney S, Momoli F, Agar M, Currow DC, Lawlor PG. The preventative role of exogenous melatonin administration to patients with advanced cancer who are at risk of delirium: study protocol for a randomized controlled trial. Trials. 2016 Aug 11;17:399. doi: 10.1186/s13063-016-1525-8. PMID 27515515
- See also: Bruyère Research Institute, Ottawa, Canada — http://www.bruyere.org/en/our-institute